CLINICAL TRIAL: NCT06073158
Title: Oesomics Anastomose Molecular Signatures of Esophageal Atresia Comparison of Biopsies Taken During the First Year of Life With Those Taken During Anastomosis
Brief Title: Molecular Signatures of Esophageal Atresia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-055; ANR (Other Grant/Funding Number: ANR-21-CE17-0042)
Record Dates: First submitted 2023-06-26; First posted 2023-10-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Atresia
Keywords: esophageal atresia; epigenetic; proteomics; metabolomics
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anastomosis group (Other): Esophageal biopsies collected during the anastomosis for the patient with esophageal atresia
  Interventions: Procedure: Esophageal biopsy collection during anastomosis
- Control group (No Intervention): Esophageal biopsies collected during a standard care endoscopy for patient with esophageal atresia during the first year of life

INTERVENTIONS:
Procedure: Esophageal biopsy collection during anastomosis — During the anastomosis, the surgeon will collect an esophageal mucosa biopsy
  Arms: Anastomosis group

SUMMARY:
Although several studies have revealed signaling pathways as well as genes potentially involved in the development of esophageal atresia (EA), our understanding of the pathophysiology of EA lags behind improvements in the surgical and clinical care of patients born with this anomaly. However, a causative genetic abnormality can be identified in less than 10% of patients, even using more recent next-generation sequencing techniques. As most cases of EA associated with tracheoesophageal fistula (TOF) are sporadic, and the familial recurrence rate is low (1%), this suggests that epigenetic and environmental factors also contribute to the disease. Further investigations are needed to better understand the mechanisms underlying EA. That information can come from the oesophageal biopsies that are collected in routine care and long-term storage at the hospital. However, the impact of the length of the storage is still unknown.

ELIGIBILITY:
Inclusion Criteria:

* Anastomosis group :

Born with esophageal atresia Anastomosis performed in Lille hospital Parents consent

- Control group : Born with esophageal atresia

Exclusion Criteria:

* Both groups :

Parents refusing to participate in the study

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the mRNA expression from esophageal biopsies between long and short term storage | The biopsies will be collected during the first year of life
  Transcriptomic profiles will be generated by the identification of mRNA and miRNA expression by 3'RNA-seq and sRNA-seq technologies. Differential expression between long and short term storage will be performed.[exploratory and untargeted analysis]
Comparison of the metabolites identification from esophageal biopsies between long and short term storage | The biopsies will be collected during the first year of life
  Metabolomic profiles will be generated (untargeted analysis that will include mnulmerous lipids, amino-acids, ...). Differential expression between long and short term storage will be performed. [exploratory and untargeted analysis]

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No